CLINICAL TRIAL: NCT02779348
Title: Effect of BIA 3-202 on the Pharmacokinetics and Pharmacodynamics of Warfarin in Healthy Volunteers
Brief Title: Effect of BIA 3-202 on the Pharmacokinetics and Pharmacodynamics of Warfarin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BIA-3202-112
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Healthy
Keywords: Nebicapone; Warfarin
MeSH Terms: interventions — nebicapone; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebicapone plus warfarin (Experimental): BIA 3-202 200 mg tid + Warfarin 25 mg
  Interventions: Drug: BIA 3-202; Drug: warfarin
- Warfarin (Experimental): Warfarin 25 mg
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: BIA 3-202 — Nebicapone tablets 200 mg
  Other Names: Nebicapone
  Arms: Nebicapone plus warfarin
Drug: warfarin — Varfine® 5 mg (warfarin 5 mg) tablets

SUMMARY:
The purpose of this study is to determine whether multiple-dose administration of nebicapone affects the pharmacokinetics of warfarin.

DETAILED DESCRIPTION:
Study design and methodology:

This was a single-centre, open-label, randomised, two-way crossover study in healthy young male and female volunteers. The study consisted of 2 treatment periods separated by a washout period of 14 days or more. In one period, subjects received nebicapone 200 mg thrice-daily (tid) for 9 days, and a warfarin 25 mg single-dose concomitantly with the morning dose of nebicapone on Day 4. In the other period, a warfarin 25 mg single-dose was administered alone. Warfarin pharmacokinetic and pharmacodynamic profiles were characterised following warfarin dosing.

ELIGIBILITY:
Inclusion Criteria:

Subjects were eligible for entry into the study if they fulfilled the following inclusion criteria:

* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Clinical laboratory test results clinically acceptable at screening and admission to first treatment period.
* Negative tests for HBsAg, anti-HCVAb and HIV-1 and HIV-2 Ab at screening.
* Negative screen for alcohol and drugs of abuse at screening and admission to each treatment period.
* Non-smokers or who smoked ≤ 10 cigarettes or equivalent per day.
* Able and willing to give written informed consent.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier, intrauterine device or abstinence.
* (If female) She had a negative urine pregnancy test at screening and admission to each treatment period.

Exclusion Criteria:

Subjects were not eligible for entry into the study if they fulfilled the following exclusion criteria:

* Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Clinically relevant surgical history.
* Personal or family history of haemostatic disorder.
* Personal or family history of bleeding complications after surgery or tooth extraction, nose or gingival bleeding, or haemorrhagic diathesis.
* Any abnormality in the coagulation tests.
* Any abnormality in the liver function tests.
* A history of relevant atopy or drug hypersensitivity.
* History of alcoholism or drug abuse.
* Consumed more than 14 units of alcohol a week.
* Significant infection or known inflammatory process at screening or admission to each treatment period.
* Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission to each treatment period.
* Had used medicines within 2 weeks of admission to first period that may affect the safety or other study assessments, in the investigator's opinion.
* Had previously received BIA 3-202.
* Had used any investigational drug or participated in any clinical trial within 6 months prior to screening.
* Had participated in more than 2 clinical trials within the 12 months prior to screening.
* Had donated or received any blood or blood products within the 3 months prior to screening.
* Vegetarians, vegans or had medical dietary restrictions.
* Cannot communicate reliably with the investigator.
* Unlikely to co-operate with the requirements of the study.
* Unwilling or unable to gave written informed consent.
* (If female) She was pregnant or breast-feeding.
* (If female) She was of childbearing potential and she did not used an approved effective contraceptive method (double-barrier, intra-uterine device or abstinence) or she used oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2006-09; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Mean Cmax of S-warfarin | before the warfarin dose, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 hours post-warfarin dose
  Maximum observed plasma drug concentration (Cmax)
Mean tmax of S-warfarin | before the warfarin dose, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 hours post-warfarin dose
  Time of occurrence of Cmax (tmax)
Mean AUC0-144 of S-warfarin | before the warfarin dose, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 hours post-warfarin dose
  Area under the plasma concentration-time curve (AUC) from time zero to 144 h post-warfarin dose (AUC0-144), calculated by the linear trapezoidal rule
Mean λz of S-warfarin | before the warfarin dose, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 hours post-warfarin dose
  Apparent terminal rate constant calculated by log-linear regression of the terminal segment of the concentration versus time curve (λz)
Mean t1/2 of S-warfarin | before the warfarin dose, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 hours post-warfarin dose
  Apparent terminal half-life, calculated from ln 2/λz (t1/2).
Mean Cmax of R-warfarin | before the warfarin dose, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 hours post-warfarin dose
  Maximum observed plasma drug concentration (Cmax)
Mean tmax of R-warfarin | before the warfarin dose, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 hours post-warfarin dose
  Time of occurrence of Cmax (tmax)
Mean AUC0-144 of R-warfarin | before the warfarin dose, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 hours post-warfarin dose
  Area under the plasma concentration-time curve (AUC) from time zero to 144 h post-warfarin dose (AUC0-144), calculated by the linear trapezoidal rule
Mean λz of R-warfarin | before the warfarin dose, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 hours post-warfarin dose
  Apparent terminal rate constant calculated by log-linear regression of the terminal segment of the concentration versus time curve (λz)
Mean t1/2 of R-warfarin | before the warfarin dose, and ½, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120 and 144 hours post-warfarin dose
  Apparent terminal half-life, calculated from ln 2/λz (t1/2).

CONTACTS AND LOCATIONS:
Locations (1):
- Human Pharmacology Unit (UFH),, S. Mamede Do Coronado, Portugal

IPD SHARING:
Plan to Share IPD: Undecided